CLINICAL TRIAL: NCT06350266
Title: Informing Low-acuity Emergency Department Patients of Non-emergent Healthcare Resources Following Discharge to Decrease Emergency Department Utilization
Brief Title: Informing Low-acuity Emergency Department Patients of Non-emergent Resources
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0183
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Emergency Service, Hospital
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Masking Description: Patients will be aware of their own messages but not of messages sent to other patients or in other arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This arm will receive no intervention outside of usual care.
- Other Healthcare Resources (Experimental): This arm will receive text messages suggesting alternatives to seeking care at a Geisinger emergency department such as seeing their Geisinger CMSL primary care provider in person or virtually (telehealth). Text suggesting these alternatives may also be included in a modified discharge paperwork packet.
  Interventions: Behavioral: Information about healthcare resources

INTERVENTIONS:
Behavioral: Information about healthcare resources — Text messages will be sent following discharge from the emergency department; text may also be modified in the (online and/or printed) discharge summary packet.
  Other Names: Text messages; Discharge summary text; Information
  Arms: Other Healthcare Resources

SUMMARY:
The goal of this campaign is to reduce unnecessary visits to a Geisinger emergency department (ED)/encourage patients with high acuity visits to follow up with an appropriate Geisinger provider. In this campaign, patients will be assigned to receive or not receive outreach following ED discharge that is aligned with the goal. Outreach will occur via a text message, as well as information added to the patient's after visit summary, and will includecalls to action to see their Geisinger CMSL PCP either in person or virtually. The study will assess whether ED use differs across patients in different outreach conditions. It will also examine whether patients follow through on the message-specific calls to action in the messages differently across conditions.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Geisinger ED visit rated as low acuity (L4 or L5)
* Discharged from Geisinger ED in past 24 hours

Exclusion Criteria:

* Cannot be contacted via the communication modality being used in the study (i.e., SMS), due to insufficient/missing contact information in the EHR or because the patient opted out
* Admitted to hospital
* Already included in intervention in past 365 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6242 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Return to Geisinger ED | within 120 days following day of discharge
  ED visit (yes/no)

OTHER OUTCOMES:
PCP appointment made | within 60 days following day of discharge
  PCP appointment made (yes/no)
PCP visit | within 60 days following day of discharge
  PCP appointment attended (yes/no)
Telehealth appointment made | within 60 days following day of discharge
  Telehealth appointment made (yes/no)
Telehealth appointment attended | within 60 days following day of discharge
  Telehealth appointment attended (yes/no)
Call made to PCP | within 60 days following day of discharge
  Record of patient call to PCP (yes/no)
Any of the suggested actions taken | within 60 days following day of discharge
  PCP called or visited, telehealth appointment attended, or PCP or telehealth appointment made (yes/no)
Urgent care visit | within 60 days following day of discharge
  Urgent care appointment attended (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT06350266/Prot_SAP_001.pdf